CLINICAL TRIAL: NCT05241873
Title: Phase I/II Study of BLU-451 in Advanced Cancers With EGFR Exon 20 Insertion Mutations
Brief Title: (Concerto) Study of BLU-451 in Advanced Cancers With EGFR Exon 20 Insertion Mutations
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision, not related to safety concerns
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BLU-451-1101
Record Dates: First submitted 2022-01-31; First posted 2022-02-16 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Lung Neoplasm Malignant; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Neoplasms; Neoplasms by Site; Lung Diseases; Respiratory Tract Disease; Carcinoma, Bronchogenic; Bronchial Neoplasms; Adenocarcinoma; Carcinoma; Neoplasms by Histologic Type; EGFR Exon 20 Mutation; EGFR Exon 20 Insertion Mutation; EGFR Activating Mutation; Antineoplastic Agents; Metastatic Lung Cancer; Brain Metastases; EGFR-mutated NSCLC; EGFR Atypical Mutations, Including G719X and L861Q
Keywords: protein kinase inhibitors; thoracic neoplasms
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Neoplasms; Neoplasms by Site; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Adenocarcinoma; Carcinoma; Neoplasms by Histologic Type; Brain Neoplasms; Thoracic Neoplasms | interventions — Carboplatin; Pemetrexed

STUDY DESIGN:
Intervention Model Description: The primary objectives of this study are in Phase 1 to identify the MTD and/or RP2D of BLU-451, and in Phase 2, to evaluate the anti-tumor activity of BLU-451.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Phase I - Part 1A Dose Escalation (Experimental): BLU-451 monotherapy with dose escalation in participants with metastatic cancer with EGFR Ex20ins or other selected EGFR mutations that have progressed after prior systemic therapies.
  Interventions: Drug: BLU-451
- Phase I - Part 1B Dose Escalation (US only) (Experimental): BLU-451 with dose escalation in combination with carboplatin and pemetrexed in participants with metastatic NSCLC with common EGFR mutations. This arm will enroll participants only in the United States.
  Interventions: Drug: BLU-451; Drug: Carboplatin; Drug: Pemetrexed
- Phase I - Part 2 BLU-451 Monotherapy Enrichment (Experimental): BLU-451 enrichment at select doses.
  Interventions: Drug: BLU-451
- Phase II - Cohort 2A (Experimental): EGFR Ex20ins participants who have previously received platinum-based chemotherapy and either amivantamab or mobocertinib will receive BLU-451.
  Interventions: Drug: BLU-451
- Phase II - Cohort 2B (Experimental): EGFR Ex20ins participants who have previously received platinum-based chemotherapy but have not received a prior EGFR Ex20ins-targeted agent will receive BLU-451.
  Interventions: Drug: BLU-451
- Phase II - Cohort 2C (Experimental): EGFR Ex20ins participants with at least one measurable lesion in brain per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 who have previously received platinum-based chemotherapy will receive BLU-451. Previous treatment with EGFR Ex20Ins-targeted therapies is allowed but not required.
  Interventions: Drug: BLU-451
- Phase II - Cohort 2D (Experimental): Participants with EGFR Ex20ins who have previously received platinum-based chemotherapy and both amivantamab AND mobocertinib, OR received any investigational Ex20Ins targeted agent(s) will receive BLU-451. Participants with Ex20ins or atypical mutations enrolled in other cohorts and who have other oncogenic drivers by central testing at baseline will be moved to this arm.
  Interventions: Drug: BLU-451
- Phase II - Cohort 2E (Experimental): Participants with EGFR Ex20ins who have not received prior systemic therapy in metastatic setting will receive BLU-451.
  Interventions: Drug: BLU-451
- Phase II - Cohort 2F (Experimental): Participants with EGFR atypical mutations (e.g., G719X, L861Q) who have previously received at least one EGFR tyrosine kinase inhibitor (TKI) will receive BLU-451. Participants with with other atypical EGFR mutations, such as S768I, may be enrolled if approved by Sponsor Medical Monitor.
  Interventions: Drug: BLU-451
- Phase II - Cohort 2G (Experimental): Participants with EGFR atypical mutations (e.g., G719X, L861Q) who have not received prior systemic therapy in metastatic setting will receive BLU-451. Participants with with other atypical EGFR mutations, such as S768I, may be enrolled if approved by Sponsor Medical Monitor.
  Interventions: Drug: BLU-451

INTERVENTIONS:
Drug: BLU-451 — BLU-451 will be administered orally by tablet QD or BID on a 21-day treatment cycle
Drug: Carboplatin — Carboplatin will be administered intravenously (IV) on Day 1 of each cycle (every 3 weeks) for 4 to 6 cycles
  Arms: Phase I - Part 1B Dose Escalation (US only)
Drug: Pemetrexed — Pemetrexed will be administered prior to carboplatin as an IV infusion on Day 1 of each cycle (every 3 weeks)
  Arms: Phase I - Part 1B Dose Escalation (US only)

SUMMARY:
This is a Phase 1/2, open-label first-in-human study of the safety, pharmacokinetics (PK), pharmacodynamics, and anti-tumor activity of BLU-451 monotherapy and BLU-451 in combination with platinum-based chemotherapy (carboplatin and pemetrexed). All participants will receive BLU-451 on a 21-day treatment cycle.

DETAILED DESCRIPTION:
The study is a Phase 1/2 Study of BLU-451 in Advanced Cancers with Epidermal growth factor receptor (EGFR) Exon 20 Insertion Mutations (Ex20ins). The study has two phases:

An initial Phase 1 portion will enroll participants with metastatic cancer with EGFR Ex20ins or other selected EGFR mutations that have progressed after prior systemic therapies and will determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of BLU-451.

Part 1B dose-escalation will enroll participants with metastatic Non-small Cell Lung Cancer (NSCLC) in the USA only to determine the MTD and/or RP2D of BLU-451 in combination with carboplatin and pemetrexed.

A Phase 2 portion will further evaluate the efficacy and safety of BLU-451 as monotherapy at RP2D in participants with NSCLC.

ELIGIBILITY:
INCLUSION CRITERIA:

All participants:

* Documented EGFR mutation, based on Next-generation sequencing (NGS) testing of tumor or liquid biopsy analyzed in a local Clinical Laboratory Improvement Amendments (CLIA) (or International Organization for Standardization (ISO) 15189)-certified or equivalent laboratory are required. Redacted copies of laboratory results must be available for Sponsor review.
* Able to provide a new or archived pretreatment formalin-fixed, paraffin-embedded (FFPE) tumor sample. For participants who received EGFR-targeted therapy subsequent to the most recent archived biopsy, all efforts should be made to obtain a new biopsy unless it is not safe or feasible to obtain one.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Participants must be without seizures for at least 14 days prior to enrollment, and patients who receive treatment with anti-epileptic drugs must be on stable doses for at least 14 days prior to enrollment.
* Adequate hematological, renal, and hepatic function:

Participants in Phase 1

* Histologically or cytologically confirmed metastatic NSCLC (stage IVA and IVB per American Joint Committee on Cancer (AJCC) 8th edition) or other metastatic cancers except for primary CNS tumors (Part 1A or Part 2 only).
* Must have evaluable or measurable disease per RECIST v1.1.
* Progression on or after or intolerance to most recent systemic therapy.

Participants in Phase 2

* Histologically or cytologically confirmed metastatic NSCLC (stage IVA and IVB per AJCC 8th edition).
* Must have measurable disease by RECIST 1.1.

EXCLUSION CRITERIA:

* Have disease that is suitable for local therapy administered with curative intent.
* Have tumor that harbors known driver alterations (including, but not limited to ROS, BRAF V600E, ALK, RET, HER2, MET, KRAS, NTRK1/2/3, EGFR C797X, or EGFR T790M mutation). These criteria are not applicable to Phase 1 Part 1B.
* Have NSCLC with mixed cell histology or a tumor with known histologic transformation (NSCLC to SCLC, SCLC to NSCLC, or epithelial to mesenchymal transition).

Other protocol-defined inclusion and exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Phase I - Determine the maximum tolerated dose (MTD) of BLU-451 | 12-15 Months
  MTD determination: Dose-limiting toxicities (DLTs) rate
Phase I - Determine the Recommended Phase 2 Dose (RP2D) of BLU-451 | 12-15 Months
  RP2D determination: DLT, PK, PD, and preliminary safety data
Phase I - Rate and severity of Adverse Events (AEs) of BLU-451 | 12-15 Months
Phase II - The Overall Response Rate (ORR) rate of BLU-451 | Up to 30 months
  ORR is defined as the proportion of subjects with objective response of CR or PR as determined by the Investigator using RECIST v1.1.

SECONDARY OUTCOMES:
Phase I - The Overall Response Rate (ORR) rate of BLU-451 | Up to 30 months
  ORR is defined as the proportion of subjects with objective response of CR or PR as determined by the Investigator using RECIST v1.1.
Phase I & II - The Duration of Response (DOR) rate of BLU-451 | 12-15 Months
  DOR is defined as the time from the first objective response (CR or PR) to documented PD per RECIST v1.1 or death within 30 days of last dose of BLU-451 from any cause.
Phase I & II - The Disease Control Rate (DCR) rate of BLU-451 | 12-15 Months
  DCR is defined as best response of CR, PR, non-CR/non-PD (for subjects who have only non-target lesions), or SD per RECIST v1.1.
Phase I & II - The Clinical Benefit Rate (CBR) of BLU-451 | 12-15 Months
  CBR is defined as confirmed response of CR or PR, or stable disease with a duration of at least 16 weeks from the first dose date.
Phase I & II - The Progression Free Survival (PFS) rate of BLU-451 | 12-15 Months
  PFS is defined as the time from the first BLU-451 dose until the date of death or the date of progression of disease or death, respectively.
Phase I & II - The Overall Survival (OS) rate of BLU-451 | 12-15 Months
  OS is defined as the time from the first BLU-451 dose until the date of death or the date of progression of disease or death, respectively.
Phase I & II - To evaluate the Central Nervous System (CNS) Overall Response Rate (ORR) of BLU-451 in subjects with measurable baseline brain metastases | Up to 30 months
  CNS ORR: Defined as the proportion of patients achieving confirmed intra-cranial CR or PR as determined by the RECIST v1.1.
Phase I & II - To evaluate the Central Nervous System (CNS) Duration of Response (DOR) of BLU-451 in subjects with measurable baseline brain metastases | Up to 30 months
  CNS DOR: Defined as the the time from the first objective intra-cranial response (CR or PR) to documented PD in patients with measurable baseline brain metastases
Phase I & II - To evaluate the Central Nervous System (CNS) Progression Free Survival (PFS) of BLU-451 in subjects with measurable baseline brain metastases | Up to 30 months
  CNS PFS: Defined as the time from the first BLU-451 dose until the date of death or the date of intra-cranial progression of disease or death, respectively in patients with measurable baseline brain metastases
Phase I - Assess treatment-induced modulation of EGFR pathway biomarkers | 12-15 Months
  Profile pharmacodynamic changes in gene expression levels of the EGFR pathway biomarkers dual specificity phosphatase (DUSP6) and sprouty RTK signaling antagonist 4 (SPRY4)
Phase I & II - To evaluate the maximum observed blood drug concentration (Cmax) of BLU-451 | Up to 30 months
Phase I & II - To evaluate the time of maximum blood concentration (tmax) of BLU-451 | Up to 30 months
Phase I & II - To evaluate the elimination half life (t1/2) of BLU-451 | Up to 30 months
Phase I & II - To evaluate the area under the blood concentration-time curve (AUC0-t, AUC0-inf) of BLU-451 | Up to 30 months
Phase I & II - To evaluate the clearance (CL/F) of BLU-451 | Up to 30 months
Phase I & II - To evaluate the volume of distribution (Vss/F) of BLU-451 | Up to 30 months
Phase II - Rate and severity of Adverse Events (AEs) of BLU-451 | Up to 30 months

CONTACTS AND LOCATIONS:
Locations (23):
- United States (13):
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - New Experimental Therapeutics of Virginia (NEXT Oncology), Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- South Korea (2):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital (CGMHLK), Taoyuan District